CLINICAL TRIAL: NCT00861497
Title: An Open-label Safety Study of Bifeprunox Investigating Flexible Doses of 20, 30, or 40mg/Day in Patients With Schizophrenia Who Have Completed Studies 10206 or 10265
Brief Title: Bifeprunox Extension to Extension Study in Patients With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study stopped after been paused (the patients were switched in the meantime)
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11051; 2005-000497-50 (EudraCT Number)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Open-label; Flexible-dose; Extension; Safety study
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bifeprunox (Experimental)
  Interventions: Drug: Bifeprunox

INTERVENTIONS:
Drug: Bifeprunox — Flexible dosage: 20, 30, or 40 mg/day

SUMMARY:
The purpose of this study is to provide access to bifeprunox for patients, who have completed previous studies with bifeprunox, and require continued treatment with bifeprunox, other treatment not being adequate. A further purpose is to investigate the safety and side-effects of bifeprunox during long-term treatment.

DETAILED DESCRIPTION:
This is a non-controlled, open-label, flexible-dose, international multi-centre extension study. The patient population consists of male and female patients with schizophrenia, who have completed open-label bifeprunox studies 10206 or 10265, and require continued treatment with bifeprunox, other treatments not being feasible as judged by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients, suffering from schizophrenia, having completed studies 10206 or 10265
* Otherwise healthy
* Female patients of non-childbearing potential, or non-pregnant, not breast-feeding women using adequate contraception
* The patient must be in need of treatment with bifeprunox (that is, the switch to another compound is not feasible)

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than schizophrenia
* Significant risk of suicide and/or violent behaviour
* Other psychiatric, neurological or behavioural disorders that may interfere with study conduct
* Substance or alcohol abuse, current cannabis dependence
* Clinically significant physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Adverse events, clinical safety laboratory tests, vital signs, ECGs, physical and neurological examinations, abnormal movement scales (AIMS, BARS, SAS) | Assessments every 4 to 8 weeks

SECONDARY OUTCOMES:
CGI-S | Assessments every 4 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- IT001, Brescia, Italy